CLINICAL TRIAL: NCT03684018
Title: Randomized Study of Two Dose Levels of Privigen in Pediatric CIDP
Brief Title: Two Dose Levels of Privigen in Pediatric CIDP
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IgPro10_4002; 2018-003430-33 (EudraCT Number)
Record Dates: First submitted 2018-09-24; First posted 2018-09-25 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Pediatric Chronic Inflammatory Demyelinating Polyneuropathy (CIDP)
MeSH Terms: interventions — Immunoglobulins, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IgPro10 (dose level 1) (Experimental)
  Interventions: Biological: IgPro10
- IgPro10 (dose level 2) (Experimental)
  Interventions: Biological: IgPro10

INTERVENTIONS:
Biological: IgPro10 — Normal human immunoglobulin G administered intravenously
  Other Names: Privigen

SUMMARY:
A randomized, open-label, prospective, multicenter study designed to investigate 2 dose levels in pediatric subjects 2 to ≤ 17 years of age with confirmed or possible CIDP, either previously exposed to IVIG treatment or unexposed to IVIG treatment

ELIGIBILITY:
Inclusion Criteria:

* - Male or female subjects 2 to ≤ 17 years of age with confirmed or possible CIDP.

Exclusion Criteria:

* - Absence of CIDP symptoms
* -History or family history of inherited neuropathy
* -Diagnosed developmental delay or regression
* -History of thrombotic episode
* -Known or suspected hypersensitivity to Privigen
* -Known allergic or other severe reactions to blood products
* -Female subject of childbearing potential either not using or not willing to use a medically reliable method of contraception or not sexually abstinent during the study
* -Pregnant or breastfeeding mother"

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2019-02-28 (Actual); Primary Completion 2029-12-20 (Estimated); Study Completion 2029-12-20 (Estimated)

PRIMARY OUTCOMES:
Percentage (%) of subjects with CIDP relapse in the Randomized Phase by dose level | Approximately 24 weeks
  CIDP relapse, defined as a clinical decline relative to the previous assessment as indicated by an increase in modified Rankin Scale (mRS) of ≥ 1 point, in the Randomized Phase

SECONDARY OUTCOMES:
Percentage of subjects with treatment emergent adverse events (TEAEs) by dose level | Approximately 56 weeks
Rate of TEAEs per infusion | Approximately 56 weeks
Rate of mild, moderate, and severe TEAEs per infusion by dose level | Approximately 56 weeks
Percentage of subjects with serious TEAEs | Approximately 56 weeks
Rate of serious TEAEs per infusion | Approximately 56 weeks
Percentage of subjects with related TEAEs | Approximately 56 weeks
Rate of related TEAEs per infusion | Approximately 56 weeks
Percentage of subjects with CIDP relapse in the Dose Exploration Phase by dose level assigned in the Randomized Phase | Approximately 24 weeks
Change in modified Rankin Scale (mRS) score from baseline in the Randomized Phase | Baseline and Approximately 24 weeks
  The mRS is a disability scale ranging from 0 (asymptomatic) to 6 (death)
Percentage (%) of subjects with CIDP improvement in the Randomization Phase by dose level | Approximately 24 weeks
  CIDP improvement in the Randomized Phase, defined as a decrease in mRS score ≥ 1 from previous visit
Percentage (%) of subjects with CIDP recovery in the Randomization Phase by dose level | Approximately 24 weeks
  CIDP recovery in the Randomized Phase, defined as decrease in mRS score as comparedto baseline AND mRS score of 1 or 0 at end of Randomized Phase
Time to CIDP relapse in Randomized Phase by dose level | Approximately 24 weeks
Percentage (%) of subjects with CIDP improvement in the Dose Exploration Phase (DEP) by dose level | Approximately 24 weeks
  CIDP improvement in the Dose Exploration Phase, defined as decrease in mRS score ≥ 1 from baseline
Percentage (%) of subjects with CIDP recovery in the Dose Exploration Phase by dose level | Approximately 24 weeks
  CIDP recovery in the Dose Exploration Phase, defined as decrease in mRS score compared to baseline AND mRS score of 1 or 0 at end of DEP
Time to CIDP Relapse in the Dose Exploration Phase by dose level | Approximately 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — CSL Behring
Locations (9):
- United States (9):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Children's Hospital of Los Angeles, Los Angeles, California
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Akron Children's Hospital, Akron, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Le Bonheur Children's Hospital, Memphis, Tennessee
  - Neurology Rare Disease Center, Denton, Texas
  - Children's Specialty Group, Norfolk, Virginia
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bus SR, de Haan RJ, Vermeulen M, van Schaik IN, Eftimov F. Intravenous immunoglobulin for chronic inflammatory demyelinating polyradiculoneuropathy. Cochrane Database Syst Rev. 2024 Feb 14;2(2):CD001797. doi: 10.1002/14651858.CD001797.pub4. PMID 38353301